CLINICAL TRIAL: NCT03005769
Title: Demographic and Clinical Predictors of Persistence in Patients Treated With Aripiprazole Once-monthly in the Italian Clinical Practice: a Retrospective Cohort, Observational Study
Brief Title: Demographic and Clinical Predictors of Persistence in Patients Treated With Aripiprazole Once-monthly in Italy
Acronym: DOMINO
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-306-00108
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia
Keywords: persistence; long-acting injectable antipsychotic; adherence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, retrospective, non-interventional study that will include schizophrenic patients who were initiated with aripiprazole once-monthly as per normal clinical practice at least 6 months before the data collection starts (inclusion visit), and is designed to evaluate demographic and clinical predictors of persistence with this treatment.

Data from each patient will be collected after informed consent is signed (inclusion visit), and will include retrospective information from the start of aripiprazole once-monthly treatment initiation (index date) until the follow-up/inclusion visit (minimum of 6 months after the index date). Data will be retrospectively collected from all visits occurring as per clinical practice (usually once monthly).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years at the time of aripiprazole once-monthly initiation)
2. Male or female
3. Diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth edition (DSM-5), available at start of aripiprazole once-monthly treatment, and confirmed by the current investigator
4. Aripiprazole once-monthly initiation (at least 1 injection) according to the clinical practice, at least 6 months before the inclusion and on June 1st 2015 or at a later date (index date)
5. Aripiprazole once-monthly was the main antipsychotic at the time of treatment initiation
6. Willingness to participate in the study; subjects must give their written consent to participate

Exclusion Criteria:

1. The patient has a psychiatric disorder other than schizophrenia as primary diagnosis
2. Participation in a clinical trial during the retrospective follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will include adult patients with schizophrenia who initiated aripiprazole once-monthly treatment as per normal clinical practice at least 6 months before data collection.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Persistence (number of days) with aripiprazole once-monthly treatment | During the first 6 months after aripiprazole once-monthly initiation.

SECONDARY OUTCOMES:
Description of aripiprazole once-monthly discontinuations and temporary interruptions and their reasons. | Through study completion, at least 6 months.
Description of health resource use related to schizophrenia (hospitalisations, outpatient visits, procedures, schizophrenia drugs) | Through study completion, at least 6 months.
Mean Clinical Global Impressions - Severity scale (CGI-S) changes | Through study completion, at least 6 months.
Characterization of the schizophrenia dimensions of the participating subjects according to the Lifetime Dimensions for Psychosis Scale (LDPS) questionnaire. | Only one time: at the end of each patient's follow-up, at least 6 months after aripiprazole once-monthly initiation
Characterization of the psychotic spectrum of the participating subjects according to Structured Clinical Interview for the Psychotic Spectrum (SCI-PSY) questionnaire. | Only one time: at the end of each patient's follow-up, at least 6 months after aripiprazole once-monthly initiation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (20):
- Italy (20):
  - Centro Salute Mentale, Ancona
  - SPDC ASST Spedali Civili, Brescia
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Policlinico "G. Rodolico", Catania
  - Policlinico Mater Domini, Catanzaro
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Casa Di Cura Neuropsichiatrica Villa Von Siebenthal, Genzano di Roma
  - Ospedale Maria S.S. dello splendore, Giulianova
  - ASL Lecce, Lecce
  - ASST Grande Ospedale Metropolitano, Milan
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Ospedale San Gerardo, Monza
  - SCDU Psichiatria. AOU San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - Clinica Psichiatrica. Università di Palermo, Palermo
  - Università degli Studi di Perugia, Perugia
  - Centro di Salute Mentale, Pomezia
  - ASL Salerno, Pontecagnano
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda ULSS 9 Treviso, Treviso

IPD SHARING:
Plan to Share IPD: No